CLINICAL TRIAL: NCT07032740
Title: Respiratory Pattern Change in Runners by Respiratory Tract Restriction Using a Respirator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Bohemia (Other)
Responsible Party: Principal Investigator, Petr Bahensky, Head of Laboratory, University of South Bohemia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: USouthBohemia
Record Dates: First submitted 2025-05-27; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Breathing Pattern
Keywords: optoelectronic plethysmography; N95; graded exercise test; abdominal compartment; chest wall compartments; FFR; face mask

STUDY DESIGN:
Intervention Model Description: Each participant underwent both tests, with and without respirators, in random order.
Who Masked: Participant
Masking Description: After enrollment in the study (in a pre-selected order of tests), participants were assigned a number under which they passed the tests.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With respirator (Experimental): The group of runners performed a test with a respirator.
  Interventions: Diagnostic Test: Bruce test
- Without respirator (Active Comparator): The group runners performed a test without a respirator.
  Interventions: Diagnostic Test: Bruce test

INTERVENTIONS:
Diagnostic Test: Bruce test — In the Bruce test, a breath pattern was obtained by means of an OEP (once with a respirator and once without a respirator).

SUMMARY:
This study involves 20 race runners (10 girls and 10 boys) aged 16-26. The investigators looked at the effect of the respirator on their respiratory function and the involvement of individual breath sectors. The order of the tests was randomly divided, each taking a test with and without a respirator.

DETAILED DESCRIPTION:
Participants in this study were race runners. The inclusion criteria required participants to be between 16 and 26 years of age, free from any injuries, and able to provide full written informed consent. Exclusion criteria included smoking or the presence of any chronic pulmonary or cardiac disease, ensuring that the study focused solely on a healthy, homogenous population of physically active individuals.

Ethical Approval Prior to the measurements, all participants signed an informed consent form. The research was carried out with the consent of the Ethics Committee, Faculty of Education, University of South Bohemia, Ref. No.: EK031/2023. All procedures performed in the study were in accordance with the ethical standards of the institutional research committee and with the Helsinki declaration.

Measures, Design and Procedures Participants visited the laboratory twice to complete GXT (graded exercise tests) with the use of OEP (pto-electronic plethysmography). The time period between testing days was 72 hours. Participants were randomly (randomizer.org) split into two groups. The first group performed tests using FFR and the second without the mask. On the second visit, participants crossed over to the other condition. The N95 respirator (Promedor24, Czech Republic) was used for the study as a gold standard in protecting against aerosol transfer during the COVID-19 pandemic. New masks were used for each test. During GXT, data from OEP were collected from the last minute of each three minute stage.

Opto-electronic plethysmography An analysis of the breathing pattern and chest wall compartment volumes was performed using opto-electronic plethysmography (BTS Bioengineering, Milan, Italy). The system involves eight cameras (five positioned anterior and three posterior to the participant) and 89 reflective markers which were placed on the subject's chest, abdomen and back in order to map the subject's trunk. This technique has been shown to be valid at rest and during maximal exercise.

The contributions of each breathing compartment (VRCp- pulmonary rib cage, VRCa- abdominal rib cage, VAb- abdomen) were determined using the difference between end-inspiratory and end-expiratory volume. The exact method of calculating chest wall kinematics with OEP has been described in prior work.

Graded Exercise Tests To complete this study, participants were asked to complete two maximal graded exercise tests (GXT) on separate days, with and without FFR. After three minutes of walking warm-up (2.7 km·h-1, 10% incline), participants completed a Bruce protocol to exhaustion (see Table 1). Bruce protocol was performed on a treadmill (Lode Valiant 2 Sport, Lode B.V., Groningen, Netherlands). All tests were carried out at the same time of day to minimize the effects of circadian rhythms.

Table 1. The number of participants in each stage of GXT. Stage Speed (km·h-1) Incline (%) Masked Unmasked

1. 2.7 10 21 21
2. 4.0 12 21 21
3. 5.4 14 20 21
4. 6.7 16 18 18
5. 8.0 18 8 13
6. 8.8 20 0 2

ELIGIBILITY:
Inclusion Criteria:

* age
* regular running training at least six times a week
* full limit for national championship

Exclusion Criteria:

* smoking
* presence of any chronic pulmonary or cardiac d

Ages: 16 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — We compare the effect of the parameter also by sex. This is determined by each participant.
Enrollment: 20 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-05-10 (Actual); Study Completion 2025-05-24 (Actual)

PRIMARY OUTCOMES:
Breathing pattern with and without using a respirator | Day 1 - first test, day 4 (after 72 hours) - second test
  Respiratory sector involvement ratio during Bruce test with using a respirator and without using a respirator

CONTACTS AND LOCATIONS:
Overall Officials: David Marko, Study Chair — University of South Bohemia in České Budějovice
Locations (1):
- University of South Bohemia, České Budějovice, Czechia

IPD SHARING:
Plan to Share IPD: Yes
The data associated with the paper are not publicly available but are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Once the article is published.
Access Criteria: If the article is in Open access mode, it will be accessible to all.

DOCUMENTS (1):
  • Informed Consent Form (2023-11-30): https://cdn.clinicaltrials.gov/large-docs/40/NCT07032740/ICF_000.pdf